CLINICAL TRIAL: NCT03863795
Title: Self-Affirmation in the Context of Stigma-Induced Identity Threat Among Smokers
Brief Title: Online Survey in Studying Smoking Attitudes and Behaviors Among Current Smokers
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCI-2019-01325; NCI-2019-01325 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-NCI-00810 (Other: NCI Division of Cancer Control and Population Sciences)
Record Dates: First submitted 2019-03-04; First posted 2019-03-05 (Actual); Results first posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Smoker

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (survey): Participants are recruited and pre-screened via an online crowdsourcing program MTurk, and then respond to a one-time research survey over 20 minutes on SurveyGizmo, an on-line survey software platform
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Respond to SurveyGizmo survey online

SUMMARY:
This trial uses an online survey to study smoking attitudes and behaviors among current smokers. An online survey consisting of questions about general demographics, smoking history, smoking attitudes, smoking behaviors, smoking intentions, health and qualities of daily life may help researchers understand the differences in smoking attitudes and behaviors among current smokers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine if self-affirmation attenuates the effects of cigarette smoking stigmatization on smoking risk perceptions, pro-smoking beliefs, and intentions to change smoking behavior.

OUTLINE:

Participants are recruited and pre-screened via an online crowdsourcing program called Amazon Mechanical Turk (MTurk). Participants then respond to a one-time research survey over 20 minutes on SurveyGizmo, an on-line survey software platform.

ELIGIBILITY:
Inclusion Criteria:

* United States (US) adult smokers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Smokers recruited through Amazon Mechanical Turk
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-03-23 (Actual); Study Completion 2019-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annette Kaufman, Principal Investigator — NCI Division of Cancer Control and Population Sciences
Locations (1):
- NCI Division of Cancer Control and Population Sciences, Rockville, Maryland, United States

REFERENCES:
- [Result] Sorgen LJ, Ferrer RA, Klein WMP, Kaufman AR. Smoking self-concept moderates the effects of self-affirmation on smoking-related beliefs and behavioral intentions. Psychol Health. 2022 Aug;37(8):964-984. doi: 10.1080/08870446.2021.1912346. Epub 2021 Apr 19. PMID 33870815

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Respondents were directed to complete a 15-20 min online survey on smoking attitudes and behaviors. Participants provided electronic informed consent and then answered two questions to confirm their current smoking status. Current established smokers (smoked at least 100 cigarettes in lifetime and now smoke every day or some days) were eligible. Eligible participants completed survey items assessing smoking characteristics and smoking self-concept.
Groups:
- Smoking Stigma, Self-Affirmation: Participants viewed a 30-s smoking stigma anti-smoking paid PSA video. Participants ranked 11 values from most to least important. Those in the self-affirmation condition wrote a short paragraph about their most important value (rank 1), describing why it was personally important and how they applied it in daily life.
- Smoking Stigma, No-Affirmation Control: Participants viewed a 30-s smoking stigma anti-smoking paid PSA video. Participants ranked 11 values from most to least important. Participants in the no-affirmation control condition wrote a short paragraph about their lowest-ranked value (rank 11), describing why it might be important to someone else.
- Non-Stigma Control, Self-Affirmation: Participants viewed a 30-s smoking non-stigma control paid PSA video. Participants ranked 11 values from most to least important. Those in the self-affirmation condition wrote a short paragraph about their most important value (rank 1), describing why it was personally important and how they applied it in daily life.
- Non-Stigma Control, No-Affirmation Control: Participants viewed a 30-s smoking non-stigma control paid PSA video. Participants ranked 11 values from most to least important. Participants in the no-affirmation control condition wrote a short paragraph about their lowest-ranked value (rank 11), describing why it might be important to someone else.
Period: Overall Study
Arm/Group | Smoking Stigma, Self-Affirmation | Smoking Stigma, No-Affirmation Control | Non-Stigma Control, Self-Affirmation | Non-Stigma Control, No-Affirmation Control
Started | 306 | 269 | 244 | 281
Completed | 306 | 269 | 244 | 281
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smoking Stigma, Self-Affirmation | Smoking Stigma, No-Affirmation Control | Non-Stigma Control, Self-Affirmation | Non-Stigma Control, No-Affirmation Control | Total
Number analyzed (Participants) | 306 | 269 | 244 | 281 | 1100
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.61 (11.201) | 37.74 (10.887) | 38.54 (11.021) | 39.70 (11.054) | 38.66 (11.054)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 121 | 101 | 96 | 118 | 436
  Female | 183 | 168 | 147 | 162 | 660
  Other | 2 | 0 | 1 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 23 | 14 | 23 | 82
  Not Hispanic or Latino | 284 | 246 | 227 | 257 | 1014
  Unknown or Not Reported | 0 | 0 | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 1 | 1 | 6
  Asian | 7 | 3 | 5 | 3 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 14 | 14 | 27 | 24 | 79
  White | 271 | 232 | 198 | 236 | 937
  More than one race | 7 | 14 | 11 | 11 | 43
  Unknown or Not Reported | 5 | 4 | 2 | 5 | 16
Region of Enrollment [Number; unit: participants]
  United States | 306 | 269 | 244 | 281 | 1100
Smoking Self-Concept [Mean (Standard Deviation); unit: units on a scale] — Smoking self-concept was assessed at baseline using the Smoking Self-Concept Scale (Shadel & Mermelstein, 1996), consisting of five items measuring smokers' agreement with statements representing a smoker self-schema. An example item is, 'Smoking is part of my personality.' Response options ranged from 1 (strongly disagree) to 5 (strongly agree). Items were averaged so that higher scores indicated a stronger smoking self-concept.
  units on a scale | 2.94 (.85) | 3.12 (.89) | 3.03 (.90) | 3.08 (.83) | 3.04 (.87)
Education [Count of Participants; unit: Participants] — Participants' education was categorized as high school graduate or less, some college, college graduate, and postgraduate.
  Participants
    High school graduate or less | 53 | 46 | 37 | 49 | 185
    Some college | 123 | 106 | 112 | 136 | 477
    College graduate | 104 | 91 | 82 | 80 | 357
    Postgraduate | 26 | 25 | 13 | 16 | 80
    Unknown | 0 | 1 | 0 | 0 | 1
Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — Nicotine dependence was assessed using the Fagerström Test for Nicotine Dependence (FTND; Heatherton et al., 1991). Six items comprise the FTND each with different point values. Points are summed to create a total score ranging from 0 to 10, with higher numbers indicating greater nicotine dependence.
  units on a scale | 4.19 (2.45) | 4.46 (2.44) | 4.53 (2.43) | 4.77 (2.49) | 4.48 (2.46)

OUTCOME MEASURES:

1. Primary Outcome: Quit Intentions
Description: Single item assessed intentions to quit smoking, 'Are you considering quitting smoking during the next 6 months?' from the 2014-2015 Tobacco Use Supplement to the Current Population Survey (1=yes, plan to stop within the next 30 days; 2=yes, plan to stop within the next 6 months, but not within 30 days; 3=no, not thinking of quitting in the next 6 months; U.S. Census Bureau, 2016). Response options were reverse scored so that higher scores indicated greater intentions to quit.
Time Frame: At the time of survey response within approximately 20 minutes
Population: Listwise deletion: 1 participant did not respond to the survey item on quit intentions. Required summary level data only. Interpretation of these unadjusted results is not recommended. Please refer to manuscript for adjusted linear regression results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smoking Stigma, Self-Affirmation | Smoking Stigma, No-Affirmation Control | Non-Stigma Control, Self-Affirmation | Non-Stigma Control, No-Affirmation Control
Number analyzed (Participants) | 306 | 269 | 244 | 280
units on a scale | 1.90 (.74) | 1.72 (.71) | 1.89 (.71) | 1.79 (.70)

2. Primary Outcome: Intentions to Switch Completely to E-cigarettes
Description: "How likely are you to switch completely from using regular cigarettes to electronic cigarettes in the next 6 months?' 1 (not at all likely) to 5 (extremely likely)
Time Frame: At the time of survey response within approximately 20 minutes
Population: Listwise Deletion: 20 participants did not respond to the intentions to switch to e-cigarettes survey item. Required summary level data only. Interpretation of these unadjusted results is not recommended. Please refer to manuscript for adjusted linear regression results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smoking Stigma, Self-Affirmation | Smoking Stigma, No-Affirmation Control | Non-Stigma Control, Self-Affirmation | Non-Stigma Control, No-Affirmation Control
Number analyzed (Participants) | 300 | 265 | 240 | 275
units on a scale | 2.29 (1.37) | 2.28 (1.44) | 2.17 (1.36) | 2.32 (1.40)

3. Primary Outcome: Intentions to Seek Cessation Counseling
Description: How likely is it that in the next 6 months you will seek counseling/support to help you quit smoking? Response options were 1 (not at all likely) to 5 (extremely likely).
Time Frame: At the time of survey response within approximately 20 minutes
Population: Listwise deletion: 28 participants did not respond to the survey item on intentions to seek cessation counseling. Required summary level data only. Interpretation of these unadjusted results is not recommended. Please refer to manuscript for adjusted linear regression results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smoking Stigma, Self-Affirmation | Smoking Stigma, No-Affirmation Control | Non-Stigma Control, Self-Affirmation | Non-Stigma Control, No-Affirmation Control
Number analyzed (Participants) | 297 | 263 | 238 | 274
units on a scale | 1.65 (1.03) | 1.60 (1.06) | 1.95 (1.25) | 1.80 (1.17)

4. Primary Outcome: Intentions to Reduce Smoking
Description: How likely is it that in the next 6 months that you will reduce the number of cigarettes you smoke in a day? Response options were 1 (not at all likely) to 5 (extremely likely).
Time Frame: At the time of survey response within approximately 20 minutes
Population: Listwise deletion: 21 participants did not respond to the survey item on intentions to reduce smoking. Required summary level data only. Interpretation of these unadjusted results is not recommended. Please refer to manuscript for adjusted linear regression results.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Smoking Stigma, Self-Affirmation | Smoking Stigma, No-Affirmation Control | Non-Stigma Control, Self-Affirmation | Non-Stigma Control, No-Affirmation Control
Number analyzed (Participants) | 303 | 262 | 240 | 274
units on a scale | 3.41 (1.32) | 3.10 (1.31) | 3.40 (1.28) | 3.19 (1.29)

5. Primary Outcome: Self-exempting Beliefs
Description: Deterministic beliefs regarding smoking behaviors were evaluated using the 18-item self-exempting beliefs scale (Oakes et al., 2004).Response options were 1 (strongly disagree) to 5 (strongly agree). Items were averaged to create a composite measure of self-exempting beliefs with excellent interitem reliability, α = .91.
Time Frame: At the time of survey response within approximately 20 minutes.
Population: Required summary level data only. Interpretation of these unadjusted results is not recommended. Please refer to manuscript for adjusted linear regression results.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smoking Stigma, Self-Affirmation | Smoking Stigma, No-Affirmation Control | Non-Stigma Control, Self-Affirmation | Non-Stigma Control, No-Affirmation Control
Number analyzed (Participants) | 306 | 269 | 244 | 281
score on a scale | 2.25 (.66) | 2.35 (.62) | 2.30 (.64) | 2.33 (.64)

6. Primary Outcome: Positive Cognitions About Smoking
Description: Five items assessed positive cognitions about smoking (Fotuhi et al., 2013). Response options were 1 (strongly disagree) to 5 (strongly agree). Items were averaged to create a composite measure of self-exempting beliefs with excellent interitem reliability, α = .91.
Time Frame: At the time of survey response within approximately 20 minutes.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Smoking Stigma, Self-Affirmation | Smoking Stigma, No-Affirmation Control | Non-Stigma Control, Self-Affirmation | Non-Stigma Control, No-Affirmation Control
Number analyzed (Participants) | 306 | 269 | 244 | 281
score on a scale | 3.15 (.76) | 3.28 (.74) | 3.25 (.80) | 3.31 (.70)

ADVERSE EVENTS:
Description: Adverse events were not monitored for this online study.
Arm/Group | Smoking Stigma, Self-Affirmation | Smoking Stigma, No-Affirmation Control | Non-Stigma Control, Self-Affirmation | Non-Stigma Control, No-Affirmation Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Required summary level data is presented per requirements. Do not interpret these unadjusted results. Please refer to the published manuscript for adjusted linear regression results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT03863795/Prot_000.pdf